CLINICAL TRIAL: NCT04861597
Title: Digital Behavioral Interventions in Inflammatory Bowel Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2021-12896; UL1TR002556 (NIH)
Record Dates: First submitted 2021-04-12; First posted 2021-04-27 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-08

CONDITIONS: Crohn Disease; Ulcerative Colitis; Inflammatory Bowel Diseases; Stress, Psychological; Depression, Anxiety
MeSH Terms: conditions — Crohn Disease; Colitis, Ulcerative; Inflammatory Bowel Diseases; Stress, Psychological; Depression; Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Internet-based cognitive behavioral therapy (Experimental): The iCBT platform selected for use in this study (Sanvello™) is an evidence-based mobile app created by clinical experts that has been shown to decrease depression, anxiety, and stress and to increase self-efficacy in a non-IBD population.15 App features include: daily mood tracking; guided journeys (e.g. psychoeducational content providing background information about cognitive behavioral therapy and instructing users on how to use app tools to maintain motivation and interest); coping tools (e.g. meditation, goal setting, and negative thought redirecting activities); weekly progress assessments; community support board.
  Interventions: Behavioral: Internet based cognitive behavioral therapy
- Digital mood tracking (Active Comparator): The digital mood tracking application (app) selected for this study (PixelTM) allows participants to log their mood each day by way of a facial expression emoji and a free-text box. This app is commercially available free of charge through iOS and Android app stores with English and Spanish language options.
  Interventions: Behavioral: Digital mood tracking

INTERVENTIONS:
Behavioral: Internet based cognitive behavioral therapy — Participants with elevated psychological distress will receive 8 weeks of internet-based cognitive behavioral therapy
  Arms: Internet-based cognitive behavioral therapy
Behavioral: Digital mood tracking — Participants with elevated psychological distress will receive 8 weeks of digital mood tracking
  Arms: Digital mood tracking

SUMMARY:
Given the bidirectionality between psychological distress and disease activity in inflammatory bowel disease (IBD), whereby increased psychological distress exacerbates disease activity and vice versa, psychosocial aspects of IBD care are receiving increased attention. However, proposed interventions are generally resource-intensive and have been tested in majority white populations. While people of color are an increasing segment of the IBD population, they are currently underrepresented in research studies. The purpose of this study is to evaluate the efficacy and implementation of internet-based cognitive behavioral therapy (iCBT) among IBD patients of color with elevated psychological distress.

DETAILED DESCRIPTION:
The investigators propose a 1:1 randomized trial design to evaluate the efficacy of iCBT among a population of Black and Latinx IBD patients and to assess factors influencing its implementation. Patients within the integrated health system at Montefiore Medical Center will be actively recruited and screened to identify those with elevated psychological distress.

Eligible patients will be randomized to receive 8 weeks of iCBT or digital mood tracking to evaluate the effect of iCBT on levels of psychological distress, HRQoL and disease activity post-intervention. The investigators will also evaluate individual process level barriers and facilitators to iCBT implementation via surveys and semi-structured interviews.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18 years
* race/ethnicity self-identified as Black/African American or Hispanic/Latino
* established diagnosis of Crohn's disease or ulcerative colitis
* elevated psychological distress: at least one T-score within two standard deviations above the mean in the domains of anxiety or depression on the National Institutes of Health Patient Reported Outcomes Measurement Information System-29 (PROMIS-29) with or without a T-score within two standard deviations above the mean for perceived stress on the National Institute of Health Toolbox Perceived Stress Scale (Perceived Stress Scale)
* internet access (smartphone/mobile device with data plan, computer with internet)
* ability to provide informed consent in English or Spanish

Exclusion Criteria:

* PROMIS-29 anxiety or depression T-scores in the severe range (above 2 standard deviations)
* Current suicidal ideation, past suicidal attempt or hospitalization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2023-03-22 (Actual); Study Completion 2023-03-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ruby Greywoode, MD, Principal Investigator — Montefiore Medical Center
Locations (1):
- Montefiore Hutchinson Campus, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gracie DJ, Guthrie EA, Hamlin PJ, Ford AC. Bi-directionality of Brain-Gut Interactions in Patients With Inflammatory Bowel Disease. Gastroenterology. 2018 May;154(6):1635-1646.e3. doi: 10.1053/j.gastro.2018.01.027. Epub 2018 Jan 31. PMID 29366841
- [Background] Mikocka-Walus A, Knowles SR, Keefer L, Graff L. Controversies Revisited: A Systematic Review of the Comorbidity of Depression and Anxiety with Inflammatory Bowel Diseases. Inflamm Bowel Dis. 2016 Mar;22(3):752-62. doi: 10.1097/MIB.0000000000000620. PMID 26841224
- [Background] Mikocka-Walus A, Bampton P, Hetzel D, Hughes P, Esterman A, Andrews JM. Cognitive-behavioural therapy has no effect on disease activity but improves quality of life in subgroups of patients with inflammatory bowel disease: a pilot randomised controlled trial. BMC Gastroenterol. 2015 May 2;15:54. doi: 10.1186/s12876-015-0278-2. PMID 25934170
- [Derived] Tiles-Sar N, Neuser J, de Sordi D, Baltes A, Preiss JC, Moser G, Timmer A. Psychological interventions for treatment of inflammatory bowel disease. Cochrane Database Syst Rev. 2025 Apr 17;4(4):CD006913. doi: 10.1002/14651858.CD006913.pub3. PMID 40243391

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 113 patients were approached at office their clinical visit. 83 patients were excluded; 37 declined to participate, 15 did not complete screening, and 31 patients were ineligible. 61 participants were consented into the study and 30 were enrolled; 18 randomized assigned to internet-Based Cognitive Behavioral Therapy arm (experimental arm), 12 randomized assigned to Digital Mood Tracking (control arm).
Groups:
- Internet-based Cognitive Behavioral Therapy (iCBT): The iCBT platform selected for use in this study (Sanvello™) is an evidence-based mobile app created by clinical experts that has been shown to decrease depression, anxiety, and stress and to increase self-efficacy in a non-inflammatory bowel disease (non-IBD) population. App features include: daily mood tracking; guided journeys (e.g. psychoeducational content providing background information about cognitive behavioral therapy and instructing users on how to use app tools to maintain motivation and interest); coping tools (e.g. meditation, goal setting, and negative thought redirecting activities); weekly progress assessments; community support board.
  Internet based cognitive behavioral therapy: Participants with elevated psychological distress will receive 4 weeks of internet-based cognitive behavioral therapy.
- Digital Mood Tracking: The digital mood tracking application (app) selected for this study (PixelTM) allows participants to log their mood each day by way of a facial expression emoji and a free-text box. This app is commercially available free of charge through iOS and Android app stores with English and Spanish language options.
  Digital mood tracking: Participants with elevated psychological distress will receive 4 weeks of digital mood tracking.
Period: Overall Study
Arm/Group | Internet-based Cognitive Behavioral Therapy (iCBT) | Digital Mood Tracking
Started | 18 | 12
Completed | 12 | 9
Not Completed | 6 | 3

BASELINE CHARACTERISTICS:
Groups:
- Internet-based Cognitive Behavioral Therapy (iCBT): The iCBT platform selected for use in this study (Sanvello™) is an evidence-based mobile app created by clinical experts that has been shown to decrease depression, anxiety, and stress and to increase self-efficacy in a non-IBD population. App features include: daily mood tracking; guided journeys (e.g. psychoeducational content providing background information about cognitive behavioral therapy and instructing users on how to use app tools to maintain motivation and interest); coping tools (e.g. meditation, goal setting, and negative thought redirecting activities); weekly progress assessments; community support board.
  Internet based cognitive behavioral therapy: Participants with elevated psychological distress will receive 4 weeks of internet-based cognitive behavioral therapy.
- Total: Total of all reporting groups
Arm/Group | Internet-based Cognitive Behavioral Therapy (iCBT) | Digital Mood Tracking | Total
Number analyzed (Participants) | 18 | 12 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 14 | 10 | 24
  >=65 years | 4 | 2 | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 8 | 19
  Male | 7 | 4 | 11
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic | 10 | 8 | 18
  Non-Hispanic Black or African American | 8 | 4 | 12
Region of Enrollment [Number; unit: participants]
  United States | 18 | 12 | 30

OUTCOME MEASURES:

1. Primary Outcome: Level of Psychological Distress
Description: Level of psychological distress in participants over the prior 7 days was measured by combining the sub-score domains of anxiety and depression from the National Institutes of Health Patient Reported Outcomes Measurement Information System-29 (PROMIS-29) assessment tool. PROMIS-29 is a 29-item form that includes 4 questions in each of the domains of anxiety and depression. Group mean scores of these 8 items are composited. Higher scores indicate a greater level of the measured trait, and raw scores are converted to a T-score that centers at a mean of 50 with a standard deviation of 10 in the general population.
Time Frame: Post-4 week trial intervention
Population: Psychological Distress data was unable to be collected for 2 participants who completed the study in the iCBT arm.
Measure: Mean (Standard Deviation); unit: T-score
Groups:
- Internet-based Cognitive Behavioral Therapy (iCBT): The iCBT platform selected for use in this study (Sanvello™) is an evidence-based mobile app created by clinical experts that has been shown to decrease depression, anxiety, and stress and to increase self-efficacy in a non-IBD population. App features include: daily mood tracking; guided journeys (e.g. psychoeducational content providing background information about cognitive behavioral therapy and instructing users on how to use app tools to maintain motivation and interest); coping tools (e.g. meditation, goal setting, and negative thought redirecting activities); weekly progress assessments; community support board.
  Internet based cognitive behavioral therapy: Participants with elevated psychological distress will receive 8 weeks of internet-based cognitive behavioral therapy
Arm/Group | Internet-based Cognitive Behavioral Therapy (iCBT) | Digital Mood Tracking
Number analyzed (Participants) | 10 | 9
T-score | 60.8 (5.6) | 59.4 (8.8)

2. Secondary Outcome: Disease Activity by Short Crohn's Disease Activity Index
Description: Disease activity over the prior 7 days for Crohn's disease patients will be measured using the Short Crohn's Disease Activity Index (sCDAI). The sCDAI consists of three variables identified as predictors of disease activity: diarrhea frequency (number of liquid or soft stools), abdominal pain, and general well-being. Scoring was calculated as follows to calculate an overall score: 44 + (2 x the number of liquid or soft stools each day for 7 days) + 5 x the sum of seven daily abdominal pain ratings (0 = none, 1 = mild, 2 = moderate, 3 = severe) + 7 x the sum of seven general well-being ratings (0 = generally well, 1 = slightly under par, 2 = poor, 3 = very poor, 4 = terrible). Overall scoring ranged from 44 to an undefined upper limit based on diarrhea frequency with increasing scores being indicative of more Crohn's disease activity. Group scores were summarized using basic descriptive statistics.
Time Frame: Post-4 week trial intervention
Population: sCDAI data was unable to be collected for 5 patients in the iCBT arm and 5 patients in the Digital Mood Tracking arm.
Measure: Mean (Standard Deviation); unit: Index Score
Groups:
- Internet-based Cognitive Behavioral Therapy (iCBT): The iCBT platform selected for use in this study (Sanvello™) is an evidence-based mobile app created by clinical experts that has been shown to decrease depression, anxiety, and stress and to increase self-efficacy in a non-IBD population. App features include: daily mood tracking; guided journeys (e.g. psychoeducational content providing background information about cognitive behavioral therapy and instructing users on how to use app tools to maintain motivation and interest); coping tools (e.g. meditation, goal setting, and negative thought redirecting activities); weekly progress assessments; community support board.
Arm/Group | Internet-based Cognitive Behavioral Therapy (iCBT) | Digital Mood Tracking
Number analyzed (Participants) | 7 | 4
Index Score | 118 (70) | 134 (69)

3. Secondary Outcome: Disease Activity by Simple Clinical Colitis Activity Index
Description: Disease activity over the prior 7 days in Ulcerative Colitis patients will be measured using the Simple Clinical Colitis Activity Index (SCCAI). The SCCAI consists of five colitis activity symptom items (bowel frequency per day, bowel frequency per night, urgency of defecation, blood in stool, and general well-being) along with an assessment of extracolonic manifestations. Bowel frequency per night is scored on a 0-2 scale and General well being is scored on a 0-4 scale. The other 3 symptom scores are scored on a 0-3 scale. 1 point each is added for the presence of any extracolonic manifestation (i.e., uveitis, pyoderma gangrenosum, erythema nodusum, and arthropathy). Scores are summarized for an overall possible scoring range of 0-19 with increasing scores being indicative of more colitis activity. Group scores were summarized using basic descriptive statistics.
Time Frame: Post-4 week trial intervention
Population: SCCAI data was unable to be collected for 75 patients in the iCBT arm and 4 patients in the Digital Mood Tracking arm.
Measure: Mean (Standard Deviation); unit: Index Score
Arm/Group | Internet-based Cognitive Behavioral Therapy (iCBT) | Digital Mood Tracking
Number analyzed (Participants) | 5 | 5
Index Score | 6 (2) | 7 (4)

4. Secondary Outcome: Perceived Stress Score
Description: Level of perceived stress in IBD patients was measured using the NIH Toolbox Item Bank/Fixed Form v2.0. This form consists of 10 questions or statements used to assess perceptions of stress in IBD patients over the past month. Responses to the 10 items are scored on a 5-point Likert scale ranging from 1 ("Never") to 5 ("Very Often"). Raw scores are auto-converted to a T-score that centers at a mean score of 50 with a Standard Deviation (SD) of 10. Higher scores are indicative of higher levels of the trait (perceived stress). Group scores were summarized using basic descriptive statistics.
Time Frame: Post-4 week trial intervention
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Internet-based Cognitive Behavioral Therapy (iCBT) | Digital Mood Tracking
Number analyzed (Participants) | 12 | 9
T-score | 58 (9) | 55 (11)

5. Secondary Outcome: Health-related Quality-of-Life
Description: Health-related Quality-of-Life as measured by the overall National Institutes of Health Patient Reported Outcomes Measurement Information System-29
Time Frame: Post-4 week trial intervention
Population: HRQoL data, other than Psychological Distress data, were not collected.
Groups:
- Internet-based Cognitive Behavioral Therapy (iCBT): The iCBT platform selected for use in this study (Sanvello™) is an evidence-based mobile app created by clinical experts that has been shown to decrease depression, anxiety, and stress and to increase self-efficacy in a non-IBD population.15 App features include: daily mood tracking; guided journeys (e.g. psychoeducational content providing background information about cognitive behavioral therapy and instructing users on how to use app tools to maintain motivation and interest); coping tools (e.g. meditation, goal setting, and negative thought redirecting activities); weekly progress assessments; community support board.
  Internet based cognitive behavioral therapy: Participants with elevated psychological distress will receive 8 weeks of internet-based cognitive behavioral therapy
Arm/Group | Internet-based Cognitive Behavioral Therapy (iCBT) | Digital Mood Tracking
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Period of trial enrollment per participants; subjects enrolled for 4 weeks, adverse event assessed post-4 week trial period.
Arm/Group | Internet-based Cognitive Behavioral Therapy (iCBT) | Digital Mood Tracking
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/12
Other Adverse Events (participants affected / at risk) | 0/18 | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-09-21): https://cdn.clinicaltrials.gov/large-docs/97/NCT04861597/Prot_SAP_000.pdf
  • Informed Consent Form (2022-09-21): https://cdn.clinicaltrials.gov/large-docs/97/NCT04861597/ICF_001.pdf